CLINICAL TRIAL: NCT03426800
Title: Acupuncture - a Treatment for Children With Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited numbers of patients
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Research Coordinator, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHN_DMK_01
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Headache
Keywords: Acupuncture; Training; Children; Effect
MeSH Terms: conditions — Headache | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Migraine_acupuncture and training (Experimental): Migraine acupuncture and training
  Interventions: Other: Acupuncture and training
- Migraine training (Experimental): Migraine training
  Interventions: Other: Acupuncture and training
- Tension_acupuncture and training (Experimental): Tension headache acupuncture and training
  Interventions: Other: Acupuncture and training
- Tension headache training (Experimental): Tension headache training
  Interventions: Other: Acupuncture and training

INTERVENTIONS:
Other: Acupuncture and training — Acupuncture twice in the week in 3 weeks combined with training in 6 weeks

SUMMARY:
Acupuncture as a treatment for headache in children

DETAILED DESCRIPTION:
A randomised controlled study in the effect of acupuncture as a treatment for headache in children.

The children are randomised for training or for training and acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by pediatrician-
* Age-9-17 years
* Min. headache 8 times within the last month

Exclusion Criteria:

* Mentally illness
* Fear of needles

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Days with headache | 30 days
  Number of days with headache

CONTACTS AND LOCATIONS:
Locations (1):
- North Denmark Hospital, Hjørring, Denmark

IPD SHARING:
Plan to Share IPD: Undecided